CLINICAL TRIAL: NCT04923451
Title: Transcranial Electrical Stimulation in Sexual Addiction: an Innovative Treatment for a Better Understanding of the Physiopathology of Craving
Brief Title: tDCS in Treatment of Craving in Sexual Addiction
Acronym: CAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier St Anne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: D20-P039
Record Dates: First submitted 2021-03-22; First posted 2021-06-11 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2020-11

CONDITIONS: Sexual Addiction; Hypersexualism
Keywords: Sexual Addiction; Hypersexualism; Neurostimulation; tDCS; fMRI
MeSH Terms: conditions — Compulsive Sexual Behavior Disorder

STUDY DESIGN:
Intervention Model Description: Quantitative data regarding the intensity of emotional response and craving to erotic images, motor inhibition task and impulsivity will be presented in the form of frequency, mean and standard deviation (SD) calculations and compared using a 2-factor repeated measures ANOVA taking into account the fact that the patient will be compared to himself (position 1 and 2 and placebo) and to other patients using 3 kinds of images (erotic, social and neutral) with 3 types of possible stimulations.
  In order to analyze the fMRI data, the regions of the patient's body will be identified. in which the BOLD activity will be correlated to the attractiveness of the image. Foreach patient, the difference before and after stimulation will be calculated. There will be no intermediate analysis.
Who Masked: Participant, Care Provider
Masking Description: Depending on the randomized group, the subject will receive one of two treatments 15 days apart (A: active anode on the right DLPFC and neutral cathode on the left shoulder; B: inactive anode on the DLPFC and inactive cathode on the left shoulder). The groups are defined as follows:
  The results of randomization will not be known by the evaluator.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patient with sexual addiction - active stimulation (Active Comparator): 25 patients with sexual addiction will be stimulated by active tDCS during 5 consecutive days
  Interventions: Device: Active Trans-cranial direct current stimulation (tDCS)
- Patient with sexual addiction - sham stimulation (placebo) (Sham Comparator): 25 patients with sexual addiction will be stimulated by sham tDCS stimulation (placebo) during 5 consecutive days
  Interventions: Device: Sham Trans-cranial direct current stimulation (tDCS)

INTERVENTIONS:
Device: Active Trans-cranial direct current stimulation (tDCS) — 5 active sessions (1/day for 5 consecutive days) of tDCS (NeuroConn DC), active anode 8cm2 on right dorso-lateral prefrontal cortex and neutral cathode, 2 mA, during 30 min will be performed
  Arms: Patient with sexual addiction - active stimulation
Device: Sham Trans-cranial direct current stimulation (tDCS) — 5 placebo sessions (1/day for 5 consecutive days) of sham tDCS (NeuroConn DC), anode 8cm2 on right dorso-lateral prefrontal cortex and neutral cathode during 30min will be performed
  Arms: Patient with sexual addiction - sham stimulation (placebo)

SUMMARY:
In patients with addiction to a substance, an increase in activity in the prefrontal cortex induced by transcranial Direct Current Stimulation -tDCS (non-invasive technique, modulating cortical activity by applying low-intensity electrical currents between two electrodes),may help reduce craving in people addicted to alcohol and tobacco. By analogy with addictive behavior with a substance, the craving observed in certain behavioral addictions would involve the same neural circuits.

The main hypothesis is to reduce the sexual craving associated with the viewing of erotic images during active brain stimulation compared to placebo stimulation. Functional MRI will allow to better understand the neural circuits involved in sexual addiction and in the expected inhibition of sexual arousal by tDCS in sexual addictions during visualization erotic images.

DETAILED DESCRIPTION:
The concept of sexual addiction appeared in American literature about 20 years ago. The term sexual addiction describes an excessive, increasing, and especially uncontrolled frequency of sexual behavior, as a conventional rule, associated with a compelling and irrepressible sexual desire (craving), which persists in spite of the possible negative consequences and personal suffering of the subject. The prevalence of this condition is estimated to be approximately 3-6% in the general population in the United States, it is independent of the socio-cultural environment. The pathophysiology of sexual addictions remains very poorly understood.

Numerous studies have focused on substance addictions and their pathophysiology. The mesolimbic dopaminergic system plays a major role in addictive behavior. The prefrontal cortex and the basolateral region of the amygdala play an important role in the craving and may cause relapse in subjects. In subjects with sexual addiction, only one controlled study has been conducted on the role of antidepressant treatment in the reduction of craving. The objective of the study is not only to evaluate the efficacy of tDCS neurostimulation in this disorder but also to identify the brain structures involved in this addictive disorder.

ELIGIBILITY:
Inclusion Criteria:

* 18-60 year old male
* Heterosexual
* Right-handed (Manual laterality test)
* With a sexual addiction (PEACCE Tool> 3 and Carnes ≥ 13/25) except for controls
* Having signed a written and informed consent
* Subject benefiting from social security

Exclusion Criteria:

* Subject presenting a medical pathology requiring drug treatment,
* Severe psychiatric pathology (bipolar disorder, hyperactivity or schizophrenia) or another addiction (alcohol, illicit substances or behavioral addiction)
* Subject consuming psychotropic drugs in progress or during the last month
* Subject not understanding French
* Subject under tutorship or curatorship
* Subjects with neurological disease including epilepsy or a history of head trauma
* Subjects hospitalized in enforced hospitalization
* Subject presenting a contraindication to tDCS: subject with an electrical or metal brain implant
* Subject with a contraindication to MRI

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2023-11-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of tDCS in treatment of craving of sexual addiction | 3 years
  The primary outcome is to assess the effectiveness of tDCS treatment on the reduction of the craving by comparing before and after active tDCS stimulation in response to erotic-pornographic images.
  Efficacy will be quantified by a sexual craving scale associated with erotico-pornographic images before and after tDCS stimulation.
  A significant decrease in craving and score on the scale is expected after tDCS stimulation. compared to control subjects. Images of social and neutral interactions will be used as comparison of expected changes.
  The scale used is the PATHOS scale: brief sexual addiction screening questionnaire.
Efficacy of tDCS in treatment of sexual addiction in subjective emotional response | 3 years
  For the evaluation of efficacy of tDCS in emotional response, indirect measurement of craving, visual emotional responses scales (Likert) will be used during visualization of erotico-pornographic images, before and after stimulation. The "desire" will be quantified on a Likert scale from 0 to 7.
Efficacy of tDCS in treatment of sexual addiction in objective emotional response | 3 years
  An assessment of emotional responses will also be done using heart rate measure during visualization of images in fMRI, before and after stimulation by tDCS

SECONDARY OUTCOMES:
Brain structures involved in sexual addiction | 3 years
  The secondary objectives are the evaluation of the brain structures involved in sexual addiction, especially craving, and the study of the modifications of the circuits involved after the application of tDCS.
  A modification of the BOLD signal in fMRI in the mesolimbic reward system as well as in the dorsolateral prefrontal cortex, orbitofrontal cortex and the amygdala in response to erotic images is expected after tDCS. 50 patients with sexual addiction will be compared with 25 healthy subjects for this objective
Evaluation of Impulsivity with The Barratt Impulsiveness Scale | 3 years
  In addition, the evaluation of impulsivity and inhibition capacities of the frontal cortex will be conducted.Changes in impulsivity scale scores and motor inhibition task scores are expected after tDCS.
Evaluation of Impulsivity with UPPS-P Impulsive Behavior Scale | 3 years
  A decrease in scores on this scale is expected after stimulation compared to patients who received placebo stimulation.
Evaluation Evaluation of Impulsivity with Stop Signal Task | 3 years
  A decrease in scores on this scale is expected after stimulation, compared to patients who received placebo stimulation.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garcia FD, Thibaut F. Sexual addictions. Am J Drug Alcohol Abuse. 2010 Sep;36(5):254-60. doi: 10.3109/00952990.2010.503823. PMID 20666699
- [Background] Malandain L, Blanc JV, Ferreri F, Thibaut F. Pharmacotherapy of Sexual Addiction. Curr Psychiatry Rep. 2020 May 7;22(6):30. doi: 10.1007/s11920-020-01153-4. PMID 32377953
- [Background] Wainberg ML, Muench F, Morgenstern J, Hollander E, Irwin TW, Parsons JT, Allen A, O'Leary A. A double-blind study of citalopram versus placebo in the treatment of compulsive sexual behaviors in gay and bisexual men. J Clin Psychiatry. 2006 Dec;67(12):1968-73. doi: 10.4088/jcp.v67n1218. PMID 17194276
- [Background] Volkow ND, Wang GJ, Fowler JS, Tomasi D, Telang F. Addiction: beyond dopamine reward circuitry. Proc Natl Acad Sci U S A. 2011 Sep 13;108(37):15037-42. doi: 10.1073/pnas.1010654108. Epub 2011 Mar 14. PMID 21402948
- [Background] Voon V, Mole TB, Banca P, Porter L, Morris L, Mitchell S, Lapa TR, Karr J, Harrison NA, Potenza MN, Irvine M. Neural correlates of sexual cue reactivity in individuals with and without compulsive sexual behaviours. PLoS One. 2014 Jul 11;9(7):e102419. doi: 10.1371/journal.pone.0102419. eCollection 2014. PMID 25013940
- [Background] Rosenberg KP, Carnes P, O'Connor S. Evaluation and treatment of sex addiction. J Sex Marital Ther. 2014;40(2):77-91. doi: 10.1080/0092623X.2012.701268. Epub 2013 Jun 21. PMID 23790248